CLINICAL TRIAL: NCT02884479
Title: An Open-Label Phase I/II Clinical Study of PT-112 in Combination With Docetaxel in Subjects With Advanced Solid Tumor in a Phase I Dose Escalation Study and in Subjects With Non-Small Cell Lung Cancer (NSCLC) in a Phase II Dose Confirmation Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SciClone Pharmaceuticals International (Cayman) Development Limited (Industry)
Collaborators: Parexel (Industry); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Organization: SciClone Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCI-PT112-ONC-P1-001
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Advanced Solid Tumor; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PT-112 + Docetaxel (Experimental): Increasing doses of intravenously administered PT-112 in combination with 60 mg/m2 docetaxel every 3 weeks (Q3W) in subjects with advanced solid tumor of any histological type.
  Interventions: Drug: PT-112; Drug: Docetaxel

INTERVENTIONS:
Drug: PT-112 — Increasing doses of intravenously administered PT-112 in combination with 60 mg/m2 docetaxel every 3 weeks (Q3W) in subjects with advanced solid tumor of any histological type.
Drug: Docetaxel — Increasing doses of intravenously administered PT-112 in combination with 60 mg/m2 docetaxel every 3 weeks (Q3W) in subjects with advanced solid tumor of any histological type.

SUMMARY:
The purpose of this study is to test PT-112 in Combination with Docetaxel in Subjects with Advanced Solid Tumor in a Phase I Dose Escalation Study and in Subjects with Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Male or female ≥ 20 years of age on the day of signing informed consent.
2. Subjects with advanced tumor of any histological type and meet the following eligibility criteria for the corresponding part of the study:

   * In Part 1, the subjects who failed at least one prior therapy must have pathologically confirmed advanced solid tumor of any histological type with preference of subjects with advanced NSCLC and either no available, or intolerable to, standard of-care treatment.
   * In Part 2, the subjects must have pathologically confirmed advanced NSCLC. Subjects are required to have evidence of measurable disease per RECIST v1.1.
3. Eastern Collaborative Oncology Group (ECOG) Performance Status ≤ 1.
4. Subject must have adequate organ function as indicated by the following laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
   * Platelets ≥ 100 × 109/L.
   * Hemoglobin ≥ 90 g/L or 5.6 mmol/L.
   * Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or calculated or directly measured creatinine clearance ≥ 60% lower limit of normal (LLN).
   * Serum total bilirubin ≤ 1.5 × ULN (subjects with Gilbert's Syndrome are allowed if direct bilirubin is within normal limits).
   * Aspartate aminotransferase (AST [SGOT]) and/or alanine aminotransferase (ALT [SGPT]) ≤ 2.5 × ULN, or ≤ 5 × ULN in presence of liver metastases.
   * International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 × ULN.
   * Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
   * Albumin ≥ 3 mg/dL.
5. Female subjects are eligible to enter and participate in the study if they are of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who
   * has had a hysterectomy
   * has had a bilateral oophorectomy (ovariectomy)
   * has had a bilateral tubal ligation
   * is post-menopausal (total cessation of menses for ≥ 1 year)
   * Childbearing potential, have a negative serum pregnancy test at screening (within 7 days of the first investigational product administration), are not breast feeding, and use adequate contraception before study entry and throughout the study until 180 days after the last investigational product administration. Adequate contraception, when used consistently and in accordance with both the product label and the instructions of the physician, are defined as follows:
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Any intra-uterine device with a documented failure rate of less than 1% per year.
   * Double barrier contraception defined as condom with spermicidal jelly, foam, suppository, or film; or diaphragm with spermicide; or male condom and diaphragm.
6. Male subjects are eligible to enter and participate in the study if they are vasectomized or agree to use of contraception during the study treatment period and for at least 180 days after the last dose of the study drug.
7. Willing and able to provide written informed consent and comply with the requirements of the study.

Exclusion Criteria:

* Subjects meeting any of the following criteria are ineligible for participation in the study:

  1. Any cytotoxic chemotherapy within 21 days, prior to initiation of study drug.
  2. Receipt of more than three prior regimens of cytotoxic chemotherapy (immunotherapy and targeted therapy will not be counted as a line of therapy).
  3. History of hypersensitivity reaction to docetaxel and polysorbate 80 or any of its components.
  4. Presence of an acute or chronic toxicity of prior chemotherapy, with the exception of alopecia, that has not resolved to Grade 1, as determined by National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03.
  5. Evidence of peripheral neuropathy of Grade 2 or greater within 28 days prior to initiation of dosing.
  6. Symptomatic brain metastasis requiring active treatment.
  7. Bone marrow reserve which, in the clinical judgment of the Principal Investigator, is not adequate for participation in this study.
  8. Known allergy or hypersensitivity to Pt-containing agents, or known intolerance to a prior Pt-containing agent which, in the judgment of the Principal Investigator, precludes re-exposure to a Pt-containing agent.
  9. Radiotherapy within 28 days prior to baseline and/or receipt of radiotherapy to >25 % of bone marrow volume.
  10. Major surgery within 28 days prior to initiation of study drug combination.
  11. Life expectancy <12 weeks.
  12. Active or clinically unstable bacterial, viral, or fungal infection requiring systemic therapy.
  13. Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
  14. Clinically significant hearing impairment, as judged by the Principal Investigator.
  15. Any of the following within 3 months prior to initiation of study drug: uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4, APPENDIX 2), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism.
  16. Unstable cardiac dysrhythmias or persistent prolongation of the QTc (Fridericia) interval to >450 msec for males or >470 msec for females.
  17. In Part 2, any previous malignancy, except for non squamous-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was successfully treated with curative intent more than two years prior to study entry.
  18. Use of any investigational agents within 28 days prior to the screening.
  19. Pregnant or lactating female.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLTs) | Day 0 to Day 28
area under the plasma concentration-time curve from 0 to the last measurable concentration (AUClast) | Cycle 1, Day 1: Pre-dose, 0.5, 1, 1.25, 1.5, 2, 3, 5, 8, 12, 24 hours post dose Cycle 1, Day 8: Pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24 hours post dose Cycle 2, Day 8: Pre-dose, 1, 2, 4 hours post dose Cycle 3 & 4, Day 8: Pre-dose

SECONDARY OUTCOMES:
Adverse Events | Cycle 1: Day 1, Day 8, Day 15; Cycle 2: Day 1, Day 8; Follow up: 30 days post final dose

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, Principal Investigator — National Cheng-Kung University Hospital
Locations (4):
- Taiwan (4):
  - Changhua Christian Hospital, Changhua County
  - China Medical University & Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes